CLINICAL TRIAL: NCT00239018
Title: A Prospective, Open-label, Multicenter, Follow-up Study on the Efficacy and Safety of Enteric-coated Mycophenolate Sodium Administered in de Novo Kidney Transplant Patients
Brief Title: Extension Study on the Efficacy and Safety of Enteric-coated Mycophenolate Sodium Administered in de Novo Kidney Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080A2405FR01E1
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: De Novo Kidney Transplantation
Keywords: Enteric-Coated Mycophenolate Sodium (EC-MPS), de novo, kidney transplantation, long-term safety.

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

SUMMARY:
The objective of this extension study is to allow patients being treated with enteric-coated mycophenolate sodium (core study CERL080A2405FR01) to continue on the same treatment and to assess the long-term safety of EC-MPS

ELIGIBILITY:
Inclusion / Exclusion Criteria

- All patients who completed study CERL080A2405-FR01 and who are willing to continue treatment with Enteric-Coated Mycophenolate Sodium.

Other protocol-defined inclusion / exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2003-04; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
To assess glomerular filtration rate at month 3 post transplantation

SECONDARY OUTCOMES:
Renal function of patients requiring post transplantation dialysis, experiencing slow graft function (defined as S. Creat level>264 μmol/l at D5) or with immediate graft function.
Incidence of patients requiring post transplantation dialysis, experience slow graft function (defined as S. Creat level>264 μmol/l at D5 or with immediate graft function.
Incidence of biopsy proven acute rejection, any treated acute rejection, and any treated acute rejection requiring antibody therapy, recurrent acute rejection and the severity of acute rejection episodes within 6 and 12 months
Incidence of graft and patient survival within 6 and 12 months
Safety and tolerability based on adverse event (AE) reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis